CLINICAL TRIAL: NCT04225910
Title: Prospective Pilot Clinical Trial of Ac225-PSMA Radioligand Therapy of Metastatic Castration-resistant Prostate Cancer
Brief Title: Clinical Trial of Ac225-PSMA Radioligand Therapy of Metastatic Castration-resistant Prostate Cancer
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XHEC-C-2019-042-2
Record Dates: First submitted 2019-10-07; First posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2019-10

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
Keywords: mCRPC, PSMA radioligand therapy, efficacy, safety
MeSH Terms: interventions — (225)Ac-PSMA-617

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mCRPC for PSMA RLT (Experimental): 225Ac-PSMA 100KBq/kg, iv. Totally 2 doses, every 8 weeks.
  Interventions: Drug: 225Ac-PSMA

INTERVENTIONS:
Drug: 225Ac-PSMA — all the patients will receive 225Ac-PSMA RLT for 2 cycles. The dosage will be calculated according to 100KBq/kg body weight. The drug will be administered by vein injection.

SUMMARY:
The death of prostate cancer patients is mainly due to metastatic castration-resistant prostate cancer. Though some new therapies has been tried to prolong the life-span of mCRPC patients, a dilemma was encountered for the drug-resistance. The PSMA RLT has been tested its efficacy and safety for the therapy of these patients. In our clinical trial, a new PSMA ligand will been used to be labeled with Ac225. This will be a prospective pilot clinical trial. 20 mCRPC patients who was incapable of 2rd ADT or chemotherapy will be recruited in this clinical tiral. The efficacy and safety of 225Ac-PSMA will be evaluated after the administration.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed prostatic adenocarcinoma.
* Clinically or imaging confirmed metastatic castration resistant prostate cancer.
* Conventional treatment failure or not available.
* PSMA avid of lesions confirmed by PSMA PET/CT.
* Hematopoietic function, kidney and liver function is normal.
* Can follow the study plan and can timely follow-up.
* Agree to sign the informed consent.

Exclusion Criteria:

* Pathological types other than the prostatic adenocarcinoma of prostate cancer.
* Not PSMA avid of lesions confirmed by PSMA PET/CT.
* Concurrent with other uncontrolled malignant tumours or five years, except for carcinoma in situ.
* Concomitant diseases are not suitable for radioactive therapy.
* Other conditions (religion, psychology, etc.) affect the informed consent, research plan, or not compliant of follow-up schedule.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-21 (Estimated)

PRIMARY OUTCOMES:
serum PSA level | through study completion, an average of 1 year
  Serum prostate specific antigen (PSA) levels was used as the main marker of efficacy evaluation, and the changes of PSA level were divided into decrease > 50%, 30% ~ 50% and < 30%.

SECONDARY OUTCOMES:
Adverse Events and Serious Adverse Events | through study completion, an average of 1 year.
  Adverse Events and Serious Adverse Events measured using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2018. CA Cancer J Clin. 2018 Jan;68(1):7-30. doi: 10.3322/caac.21442. Epub 2018 Jan 4. PMID 29313949
- [Background] Patrikidou A, Loriot Y, Eymard JC, Albiges L, Massard C, Ileana E, Di Palma M, Escudier B, Fizazi K. Who dies from prostate cancer? Prostate Cancer Prostatic Dis. 2014 Dec;17(4):348-52. doi: 10.1038/pcan.2014.35. Epub 2014 Oct 14. PMID 25311767
- [Background] Gillessen S, Omlin A, Attard G, de Bono JS, Efstathiou E, Fizazi K, Halabi S, Nelson PS, Sartor O, Smith MR, Soule HR, Akaza H, Beer TM, Beltran H, Chinnaiyan AM, Daugaard G, Davis ID, De Santis M, Drake CG, Eeles RA, Fanti S, Gleave ME, Heidenreich A, Hussain M, James ND, Lecouvet FE, Logothetis CJ, Mastris K, Nilsson S, Oh WK, Olmos D, Padhani AR, Parker C, Rubin MA, Schalken JA, Scher HI, Sella A, Shore ND, Small EJ, Sternberg CN, Suzuki H, Sweeney CJ, Tannock IF, Tombal B. Management of patients with advanced prostate cancer: recommendations of the St Gallen Advanced Prostate Cancer Consensus Conference (APCCC) 2015. Ann Oncol. 2015 Aug;26(8):1589-604. doi: 10.1093/annonc/mdv257. Epub 2015 Jun 3. PMID 26041764
- [Background] Asselah J, Sperlich C. Post-docetaxel options for further survival benefit in metastatic castration-resistant prostate cancer: Questions of choice. Can Urol Assoc J. 2013 Jan-Feb;7(1-2 Suppl 1):S11-7. doi: 10.5489/cuaj.274. PMID 23682301
- [Background] Tannock IF, de Wit R, Berry WR, Horti J, Pluzanska A, Chi KN, Oudard S, Theodore C, James ND, Turesson I, Rosenthal MA, Eisenberger MA; TAX 327 Investigators. Docetaxel plus prednisone or mitoxantrone plus prednisone for advanced prostate cancer. N Engl J Med. 2004 Oct 7;351(15):1502-12. doi: 10.1056/NEJMoa040720. PMID 15470213
- [Background] Berthold DR, Pond GR, Soban F, de Wit R, Eisenberger M, Tannock IF. Docetaxel plus prednisone or mitoxantrone plus prednisone for advanced prostate cancer: updated survival in the TAX 327 study. J Clin Oncol. 2008 Jan 10;26(2):242-5. doi: 10.1200/JCO.2007.12.4008. PMID 18182665
- [Background] de Bono JS, Oudard S, Ozguroglu M, Hansen S, Machiels JP, Kocak I, Gravis G, Bodrogi I, Mackenzie MJ, Shen L, Roessner M, Gupta S, Sartor AO; TROPIC Investigators. Prednisone plus cabazitaxel or mitoxantrone for metastatic castration-resistant prostate cancer progressing after docetaxel treatment: a randomised open-label trial. Lancet. 2010 Oct 2;376(9747):1147-54. doi: 10.1016/S0140-6736(10)61389-X. PMID 20888992
- [Background] de Bono JS, Logothetis CJ, Molina A, Fizazi K, North S, Chu L, Chi KN, Jones RJ, Goodman OB Jr, Saad F, Staffurth JN, Mainwaring P, Harland S, Flaig TW, Hutson TE, Cheng T, Patterson H, Hainsworth JD, Ryan CJ, Sternberg CN, Ellard SL, Flechon A, Saleh M, Scholz M, Efstathiou E, Zivi A, Bianchini D, Loriot Y, Chieffo N, Kheoh T, Haqq CM, Scher HI; COU-AA-301 Investigators. Abiraterone and increased survival in metastatic prostate cancer. N Engl J Med. 2011 May 26;364(21):1995-2005. doi: 10.1056/NEJMoa1014618. PMID 21612468
- [Background] Scher HI, Fizazi K, Saad F, Taplin ME, Sternberg CN, Miller K, de Wit R, Mulders P, Chi KN, Shore ND, Armstrong AJ, Flaig TW, Flechon A, Mainwaring P, Fleming M, Hainsworth JD, Hirmand M, Selby B, Seely L, de Bono JS; AFFIRM Investigators. Increased survival with enzalutamide in prostate cancer after chemotherapy. N Engl J Med. 2012 Sep 27;367(13):1187-97. doi: 10.1056/NEJMoa1207506. Epub 2012 Aug 15. PMID 22894553
- [Background] Sartor O, Coleman R, Nilsson S, Heinrich D, Helle SI, O'Sullivan JM, Fossa SD, Chodacki A, Wiechno P, Logue J, Widmark A, Johannessen DC, Hoskin P, James ND, Solberg A, Syndikus I, Vogelzang NJ, O'Bryan-Tear CG, Shan M, Bruland OS, Parker C. Effect of radium-223 dichloride on symptomatic skeletal events in patients with castration-resistant prostate cancer and bone metastases: results from a phase 3, double-blind, randomised trial. Lancet Oncol. 2014 Jun;15(7):738-46. doi: 10.1016/S1470-2045(14)70183-4. Epub 2014 May 13. PMID 24836273
- [Background] Kantoff PW, Higano CS, Shore ND, Berger ER, Small EJ, Penson DF, Redfern CH, Ferrari AC, Dreicer R, Sims RB, Xu Y, Frohlich MW, Schellhammer PF; IMPACT Study Investigators. Sipuleucel-T immunotherapy for castration-resistant prostate cancer. N Engl J Med. 2010 Jul 29;363(5):411-22. doi: 10.1056/NEJMoa1001294. PMID 20818862
- [Background] Summers N, Vanderpuye-Orgle J, Reinhart M, Gallagher M, Sartor O. Efficacy and safety of post-docetaxel therapies in metastatic castration-resistant prostate cancer: a systematic review of the literature. Curr Med Res Opin. 2017 Nov;33(11):1995-2008. doi: 10.1080/03007995.2017.1341869. Epub 2017 Jul 10. PMID 28604117
- [Background] Kopka K, Benesova M, Barinka C, Haberkorn U, Babich J. Glu-Ureido-Based Inhibitors of Prostate-Specific Membrane Antigen: Lessons Learned During the Development of a Novel Class of Low-Molecular-Weight Theranostic Radiotracers. J Nucl Med. 2017 Sep;58(Suppl 2):17S-26S. doi: 10.2967/jnumed.116.186775. PMID 28864607
- [Background] Allen BJ. A comparative evaluation of Ac225 vs Bi213 as therapeutic radioisotopes for targeted alpha therapy for cancer. Australas Phys Eng Sci Med. 2017 Jun;40(2):369-376. doi: 10.1007/s13246-017-0534-6. Epub 2017 Mar 24. PMID 28342027
- [Background] Kratochwil C, Bruchertseifer F, Rathke H, Bronzel M, Apostolidis C, Weichert W, Haberkorn U, Giesel FL, Morgenstern A. Targeted alpha-Therapy of Metastatic Castration-Resistant Prostate Cancer with 225Ac-PSMA-617: Dosimetry Estimate and Empiric Dose Finding. J Nucl Med. 2017 Oct;58(10):1624-1631. doi: 10.2967/jnumed.117.191395. Epub 2017 Apr 13. PMID 28408529